CLINICAL TRIAL: NCT05644470
Title: Association of Implant Position and Crown Contour With Esthetics and Tissue Health in Anterior Single Tooth Replacement: a Prospective Study
Brief Title: Association of Implant Position and Crown Contour With Tissue Health
Status: Recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Chief professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: SH9H-2022-T296
Record Dates: First submitted 2022-11-26; First posted 2022-12-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Dental Implants
Keywords: dental implants; emergence profile; crown contour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Peri-implant crevicular fluid will be collected to analyze the inflammatory cytokine. Sub-mucosal plaque will be collected to analyze the composition of microbiome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental implant rehabilitation: Patients having undergone dental implant treatment, with a single implant-supported restoration in anterior jaws (premolars to premolars), will be included.

SUMMARY:
Emergence profile and crown contour of implant supported rehabilitation, which is influenced by implant position, is associated with peri-implant health and esthetic outcomes. However, there is no study prospectively explore the association between implant position, emergence profile/crown contour, and dental implant outcomes. Thus, the present study aims to (1) assess the multivariate association between local factors and peri-implant soft-tissue health, inflammation, and microbiome; and (2) to identify patterns/clusters of implant characteristics significantly associated with health or inflammation.

DETAILED DESCRIPTION:
This will be a prospective study aimed at associating the development of peri-implant mucosal inflammation (mucositis) and deeper inflammation (peri-implantitis with marginal bone loss) with features associated with implant position (three-dimensional position of the implant platform) and the consequent shape of the crown contour and emergence profile. The hypothesis is that implant position determines the shape of the crown, which in turn determines the persistence of a local microbial biofilm as unfavourable crown contours hamper oral hygiene efforts aimed at biofilm control/removal. The persistence of a biofilm will cause soft tissue inflammation, which may lead to microbial dysbiosis and disease.

ELIGIBILITY:
Inclusion Criteria:

Patients with a single implant-supported restoration in anterior jaws (premolars to premolars), with adjacent natural teeth, with pre-surgery CBCT and intra-oral scans, and willing to comply with research appointments/schedule.

Exclusion Criteria:

* Pregnancy or intention to become pregnant at any point during the study duration;
* With any systematic diseases/conditions that are contradictions to dental implant treatment;
* Inability or unwillingness of individual to give written informed consent.
* Inability of follow-up according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will have undergone pre-surgery examination (including CBCT and intra-oral scan) received dental implant treatment in Department of Oral Implantology, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine. Timing of implant placement will be type 3/4. Patients will have one single implant supported rehabilitation in anterior jaws (premolar to premolar), with adjacent natural teeth.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in bleeding on probing | Changes over six months, 1, 2, and 3 years after final crown insertion.
  Peri-implant probing will be performed with light (∼25 g) force using UNC-15 periodontal probe, at six sites (mesio- buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) per implant. At each site, presence of bleeding will be recorded.

SECONDARY OUTCOMES:
Changes in cytokine level in peri-implant crevicular fluid | Changes over six months, 1, 2, and 3 years after final crown insertion.
  Peri-implant crevicular fluid will be collected and level of inflammatory cytokines will be analyzed using commercial enzyme-linked immunosorbent assays (ELISAs) kits.
Changes in composition of microbiome in sub-gingival plaque sample | Changes over six months, 1, 2, and 3 years after final crown insertion.
  Sub-gingival plaque sample will be collected. Composition of microbiome in sub-gingival plaque samples will be assessed by 16sRNA technique.
Marginal bone level change | Chenges over Six months, 1, 2, and 3 years after final crown insertion.
  Marginal bone level change will be measured on periapical radiograph using parallel technique. The uppermost end of bone-to-implant contact will be recorded as marginal bone level. Implant will be used as reference.
Buccal soft tissue level change | Changes over six months, 1, 2, and 3 years after final crown insertion.
  Intra-oral scan taken at different follow-up time points will be superimposed. Buccal soft tissue level will be recorded and the change will be measured.
Papilla height change | Changes over six months, 1, 2, and 3 years after final crown insertion.
  Intra-oral scan taken at different follow-up time points will be superimposed. Papilla height will be recorded and the change will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD, Principal Investigator — Shanghai Ninth People Hospital
Locations (1):
- Department of Oral and Maxillo-facial Implantology, Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katafuchi M, Weinstein BF, Leroux BG, Chen YW, Daubert DM. Restoration contour is a risk indicator for peri-implantitis: A cross-sectional radiographic analysis. J Clin Periodontol. 2018 Feb;45(2):225-232. doi: 10.1111/jcpe.12829. Epub 2017 Dec 5. PMID 28985447
- [Background] Yi Y, Koo KT, Schwarz F, Ben Amara H, Heo SJ. Association of prosthetic features and peri-implantitis: A cross-sectional study. J Clin Periodontol. 2020 Mar;47(3):392-403. doi: 10.1111/jcpe.13251. Epub 2020 Jan 21. PMID 31912511
- [Background] Chan D, Pelekos G, Ho D, Cortellini P, Tonetti MS. The depth of the implant mucosal tunnel modifies the development and resolution of experimental peri-implant mucositis: A case-control study. J Clin Periodontol. 2019 Feb;46(2):248-255. doi: 10.1111/jcpe.13066. Epub 2019 Feb 7. PMID 30638273
- [Background] Tonetti MS, Jung RE, Avila-Ortiz G, Blanco J, Cosyn J, Fickl S, Figuero E, Goldstein M, Graziani F, Madianos P, Molina A, Nart J, Salvi GE, Sanz-Martin I, Thoma D, Van Assche N, Vignoletti F. Management of the extraction socket and timing of implant placement: Consensus report and clinical recommendations of group 3 of the XV European Workshop in Periodontology. J Clin Periodontol. 2019 Jun;46 Suppl 21:183-194. doi: 10.1111/jcpe.13131. PMID 31215112